CLINICAL TRIAL: NCT01561664
Title: Relations Between Obesity and Insulin Resistance: Role of Inflammation Regulatory Mechanisms in Obese Patients Without Associated Comorbidity
Brief Title: Inflammation Regulation in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 8685
Record Dates: First submitted 2012-03-06; First posted 2012-03-23 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2012-03

CONDITIONS: Obesity; Insulin Resistance
Keywords: obesity; insulin resistance
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- volunteers (Active Comparator): not overweight Volunteers responding to the study criteria
  Interventions: Other: muscle and fat biopsy
- overweight patients insulin sensitive (Experimental): overweight patients insulin sensitive responding to the study criteria
  Interventions: Other: muscle and fat biopsy
- overweight insulin resistant (Experimental): overweight patients insulin resistant responding to the study criteria
  Interventions: Other: muscle and fat biopsy

INTERVENTIONS:
Other: muscle and fat biopsy — muscle and fat biopsy

SUMMARY:
Insulin resistance is one of the main mechanisms involved in metabolic diseases. inflammation has been implicated in its pathogenesis, due to innate immunity activation by free fatty acids, lipopolysaccharides (LPS) and lactate. Free fatty acids, LPS and lactate activate innate immunity in squelettal muscle and adipose tissue via Toll-like receptor 2/4, NFkB, IRF3 (Interferon Responsive Factor 3) and cytokines secretion (TNFa, IFN g, IL1b, IL6), chemokines secretion (MCP1) and leukotrienes (LTB4). Feed back mechanisms involved in TLR signaling pathways as RLI (ribonuclease L inhibitor)/ABCE1, have never been studied in inflammation due to obesity. RLI inhibits an endoribonuclease, RNase L, which has been recently implicated in TLR signaling The purpose of this study is to analyse the role of RLI and RNase L in TLR regulation, and its potential implication in the link between obesity, inflammation and insulin resistance in adipose tissue and squeletal muscle in humans.

DETAILED DESCRIPTION:
The investigators working hypothesis is that RNase L and RLI contribute to chronic inflammation regulation and to insulin response through TLR 4 pathway regulation in obesity. The investigators main purpose is to compare innate immunity activation pathway between insulin sensitive, insulin resistant obese patients and control patients. Insulin sensitive and insulin resistant obese patients will be distinguish thanks to the HOMA ir index. The investigators second objectives are to evaluate if the degree of inflammation in adipose tissue and squeletal muscle is correlated to insulin sensitivity measured by hyperinsulinemic euglycemic clamp and to characterise inflammatory pathway and regulation pathway. A special focus will be given to the leukotrienes and their potential role in insulin resistance pathogenesis. The investigators will have two approaches:- characterisation of subjects with normal weight, of obese insulin sensitive and obese insulin resistant through a metabolic evaluation, an inflammatory characterisation and a measure of insulin sensitivity at the systemic level, in adipose tissue and in squeletal muscle.- an in vitron approach with human myoblast and adipocytes culture, extracted from the investigators patients: characterisation of inflammation, innate immunity.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 65 years old
* Men/ menopausal women
* BMI <25 kg/m2 for the control group, BMI >30 kg/m2 for the obese group
* Non diabetic patients
* HOMAIR <3 for the insulin sensitive obese group
* Non smoking
* Without any inflammatory disease
* Without any first degrees relative with diabetes
* Without any treatment that could interfere with insulin sensitivity
* without any infection

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-11; Primary Completion 2011-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
TLR regulation | 2 years
  analyse the role of RLI and RNase L in TLR regulation, and its potential implication in the link between obesity, microinflammation and insulin resistance in adipose tissue and squelettal muscle in humans.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Mercier, Study Chair — University Hospital, Montpellier
Locations (1):
- Montpellier University Hospital, Montpellier, France